CLINICAL TRIAL: NCT04804527
Title: Intensified In-hospital Physiotherapy for Patients After Hip Fracture Surgery (IPPAHS). A Pragmatic, Randomized Feasibility Trial.
Brief Title: Intensified In-hospital Physiotherapy for Patients After Hip Fracture Surgery.
Acronym: IPPAHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Gigtforeningen (Other); Danske Fysioterapeuter (Other)
Responsible Party: Principal Investigator, Theresa Bieler, Research Therapist, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2020-828
Record Dates: First submitted 2021-03-04; First posted 2021-03-18 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Hip Fractures
Keywords: Exercise Therapy; Physical Therapy Modalities; Mobility Limitation; Feasibility Studies
MeSH Terms: conditions — Hip Fractures; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, randomized, controlled, unblinded feasibility trial with two parallel groups: an intervention group receiving intensified acute in-hospital physiotherapy (n=40) and a control group receiving usual care acute in-hospital physiotherapy (n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensified physiotherapy (Experimental): In addition to usual care physiotherapy patients in the intensified physiotherapy group will receive an extra physiotherapy session of up to 30 minutes on every weekday starting on the first postoperative day. The session will include progressive functional training of basic mobility and walking in the ward delivered by an experienced physiotherapist affiliated with the trial. The aim of this additional session is to improve the functional advances achieved during the earlier physiotherapy session.
  Interventions: Other: Intensified physiotherapy
- Usual care physiotherapy (Active Comparator): Patients will receive approximately 30 minutes physiotherapy once daily in the ward delivered by the ward's usual physiotherapists i.e. starting on the first postoperative day and thereafter primarily on weekdays until discharge (a mean of 8.82 days after admission). Usual care physiotherapy is individualized taking the patients ability and previous level of functioning into account and includes 1) progressive functional training of basic mobility e.g. in-out of bed, sit-to-stand and walking including progression in walking aid, stair training if possible, and advices toward better physical functional level, 2) basic bed exercises with progression to standing exercises according to a hand-out training program and recommendations on doing exercises daily and being as physical active as possible during the day.
  Interventions: Other: Usual care physiotherapy

INTERVENTIONS:
Other: Intensified physiotherapy — Physiotherapy x2
  Arms: Intensified physiotherapy
Other: Usual care physiotherapy — Physiotherapy x1
  Arms: Usual care physiotherapy

SUMMARY:
Regaining basis mobility after a hip fracture surgery is an important in-hospital rehabilitation goal because patients who have regained basis mobility at pre-fracture level at discharge have lower 30-day mortality and readmission rate and are more likely to be discharged to their own home. However, at discharge only half of the patients have regained their pre-fracture basis mobility level.

Intensified acute in-hospital physiotherapy (e.g. more than once daily) highlighting weight-bearing activities and ambulation could have a positive effect on the proportion of patients who regain their pre-facture basic mobility at discharge. However, data from daily clinical practice suggest that only half of the patients are able to complete physiotherapy on the first postoperative day and that fatigue, hip fracture-related pain and habitual cognitive status are the most frequent reasons for not completing planned physiotherapy (once daily) during the first three postoperative days. Thus to undertake an RCT investigating the effect of intensified acute in-hospital physiotherapy i.e. two daily sessions of physiotherapy compared to usual care i.e. one daily session, on regained pre-facture basic mobility at discharge in patients with hip fracture raises important practical concerns regarding e.g. completion rate of planned physiotherapy. The potential positive effects of intensified physiotherapy will be hampered if too many patients are unable to complete planned physiotherapy e.g. because of fatigue or pain. Feasibility studies ask whether something can be done and are preliminary studies conducted specifically for the purposes of establishing whether or not a full trial will be feasible to conduct. Thus, the main aim of the trial is to assess the feasibility of conducting a definitive pragmatic RCT in terms of implementation, practicality and acceptability of intensified acute in-hospital physiotherapy i.e. two daily sessions of physiotherapy highlighting weight-bearing activities and ambulation on weekdays among patients with hip fracture.

The main predefined feasibility criterium is that about twice as many physiotherapy sessions are completed in the intensified physiotherapy group compared to in the usual care physiotherapy group.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if he/she meets the following criteria:

* Diagnosed with an isolated, first time hip fracture on the affected side
* Age ≥ 65 years
* Able to speak and understand Danish
* Home-dwelling with an independent pre-fracture ability to walk indoors (New Mobility Score (NMS) ≥ 2)
* Able to give written informed consent prior to physiotherapy in the first postoperative day

Exclusion Criteria:

A participant will be excluded from the study if he/she meets any of the following criteria:

* The fracture is pathological (e.g. cancer-based)
* Postoperative weight-bearing is restricted
* Multiple body fractures are present
* Serious postoperative medical complications occur
* Any other conditions that in the opinion of the investigator makes a potential participant unfit for participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Total physiotherapy completion rate during hospitalization | Through hospital stay, an average of 8.82 days after admission.
  The degree of completion (successful completion, partial completion or cancellation) of every physiotherapy session on weekdays from the first postoperative day to discharge will be rated by the physiotherapists and total physiotherapy completion rate during hospitalization will be calculated. The physiotherapists will also register cause of partial completion or cancellation.

SECONDARY OUTCOMES:
Hip-fracture-related pain at rest | Through hospital stay, an average of 8.82 days after admission.
  Measured at rest before physiotherapy using a five-point (no, slight, moderate, severe, unbearable pain) Verbal Rating Scale (VRS) on weekdays from the first postoperative day to discharge.
Hip-fracture-related pain during physiotherapy | Through hospital stay, an average of 8.82 days after admission.
  Measured during physiotherapy using a five-point (no, slight, moderate, severe, unbearable pain) Verbal Rating Scale (VRS) on weekdays from the first postoperative day to discharge.
Fatigue at rest | Through hospital stay, an average of 8.82 days after admission.
  Measured at rest before physiotherapy using a five-point (no, slight, moderate, severe, unbearable fatigue) Verbal Rating Scale (VRS) on weekdays from the first postoperative day to discharge.
Fatigue during physiotherapy | Through hospital stay, an average of 8.82 days after admission.
  Measured during physiotherapy using a five-point (no, slight, moderate, severe, unbearable fatigue) Verbal Rating Scale (VRS) on weekdays from the first postoperative day to discharge.
Upright time during hospitalization | From the second postoperative day to discharge, though for a maximum of 10 days after surgery.
  Time spend standing or walking assessed by using a body-worn accelerometer-based activity monitor (ActivePAL3c). The monitor will be attached to the thigh of the non-operated leg on the first postoperative day and the patient will wear the monitor continuously during hospitalization.
Upright events during hospitalization | From the second postoperative day to discharge, though for a maximum of 10 days after surgery.
  Transitions from sitting to standing assessed by using a body-worn accelerometer-based activity monitor (ActivePAL3c). The monitor will be attached to the thigh of the non-operated leg on the first postoperative day and the patient will wear the monitor continuously during hospitalization.
Basic mobility assessed using The Cumulated Ambulation Score (CAS) | Through hospital stay, an average of 8.82 days after admission.
  Basic mobility measured by using the Cumulated Ambulation Score (CAS) will be assessed in conjunction with every physiotherapy session on weekdays from the first postoperative day to discharge. The CAS is a tester administered score which describes the patient's independency in (1) getting in and out of bed, (2) sit to stand from a chair, and (3) walking ability (with and without walking aid). Each activity is assessed on a three-point ordinal scale from 0 to 2 (0: Not able to with human assistance and verbal cueing, 1: able to with human assistance or verbal cueing 2: Able to safely without human assistance or verbal cueing) resulting in a total CAS score between 0 and 6 (6 indicating independent ambulation).
Regain of pre-fracture basic mobility level at discharge | Baseline (pre-fracture) and at discharge an average of 8.82 days after admission
  Basic mobility measured by using the Cumulated Ambulation Score (CAS). The CAS is a tester administered score which describes the patient's independency in (1) getting in and out of bed, (2) sit to stand from a chair, and (3) walking ability (with and without walking aid). Each activity is assessed on a three-point ordinal scale from 0 to 2 (0: Not able to with human assistance and verbal cueing, 1: able to with human assistance or verbal cueing 2: Able to safely without human assistance or verbal cueing) resulting in a total CAS score between 0 and 6 (6 indicating independent ambulation).

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Bieler, PhD, Study Director — Bispebjerg and Frederiksberg Hospital, Dept. of Physical & Occupational Therapy
Locations (1):
- Bispebjerg Hospital, Department of Physical & Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No